CLINICAL TRIAL: NCT00535925
Title: Nephropathy in Type 2 Diabetes: Effects of an Intensive Multifactorial Intervention Trial on Cardio-renal Events.
Brief Title: Nephropathy In Type 2 Diabetes and Cardio-renal Events
Acronym: NID-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Ferdinando Carlo Sasso, MD, PhD, AssociateProfessor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 246813579
Record Dates: First submitted 2007-09-24; First posted 2007-09-27 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Nephropathy
Keywords: type 2 diabetes; nephropathy; cardiovascular (CV) events
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Kidney Diseases | interventions — Irbesartan; Ramipril; Hydrochlorothiazide; Furosemide; Amlodipine; Atenolol; Doxazosin; Clonidine; Insulin; Simvastatin; Fibric Acids; Erythropoietin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (SoC) therapy (Active Comparator): Control group patients will continue their SoC therapy. During the study such patients could receive all the therapeutic modifications according to the good medical practice of the specialist.
  Interventions: Drug: SoC therapy
- Multifactorial Intensified therapy (Experimental): An intensive multifactorial intervention according Scientific Guidelines is performed to achieve the goals for the following risk factors: hypertension, hyperglycaemia, lipids, anaemia.
  In particular, new antihypertensive drugs will be added one by one until the achievement of blood pressure target (<130/80 mmHg).
  Interventions: Drug: irbesartan; Drug: ramipril; Drug: hydrochlorothiazide; Drug: furosemide; Drug: amlodipine; Drug: atenolol; Drug: doxazosin; Drug: clonidine; Drug: insulin; Drug: simvastatin; Drug: fibrate; Drug: erythropoietin; Drug: aspirin

INTERVENTIONS:
Drug: SoC therapy — the patients have to be treated according the standard good medical practice by any center
  Arms: Standard of Care (SoC) therapy
Drug: irbesartan — Therapy for hypertension:
  - Step 1: irbesartan 300 mg/die and ramipril 10 mg/die
  Arms: Multifactorial Intensified therapy
Drug: ramipril — Therapy for hypertension:
  - Step 1: irbesartan 300 mg/die and ramipril 10 mg/die
  Arms: Multifactorial Intensified therapy
Drug: hydrochlorothiazide — Therapy for hypertension
  - Step 2: Diuretic (hydrochlorothiazide 12.5-25 mg/die if serum creatinine <2 mg/dl, furosemide 25-75 mg/die if serum creatinin ≥2 mg/dl)
  Arms: Multifactorial Intensified therapy
Drug: furosemide — Therapy for hypertension
  - Step 2: Diuretic (hydrochlorothiazide 12.5-25 mg/die if serum creatinine <2 mg/dl, furosemide 25-75 mg/die if serum creatinin ≥2 mg/dl)
  Arms: Multifactorial Intensified therapy
Drug: amlodipine — Therapy for hypertension
  - Step 3: amlodipine up to 10 mg/die
  Arms: Multifactorial Intensified therapy
Drug: atenolol — Therapy for hypertension
  - Step 4: atenolol up to 100 mg/die
  Arms: Multifactorial Intensified therapy
Drug: doxazosin — Therapy for hypertension
  - Step 5: doxazosin up to 4 mg/die
  Arms: Multifactorial Intensified therapy
Drug: clonidine — Therapy for hypertension
  - Step 6: clonidine
  Arms: Multifactorial Intensified therapy
Drug: insulin — Therapy for Hyperglycaemia (to achieve HbA1c <7):
  - insulin
  Arms: Multifactorial Intensified therapy
Drug: simvastatin — Therapy for hypercholesterolemia:
  - for reducing LDL cholesterol < 100 mg/dl: simvastatin up to 80 mg/die
  Arms: Multifactorial Intensified therapy
Drug: fibrate — Therapy for hypertriglyceridemia
  - for reducing triglycerides < 150 mg/dl and/or increasing HDL cholesterol > 40-50 mg/dl: a fibrate
  Arms: Multifactorial Intensified therapy
Drug: erythropoietin — Treatment of anaemia:
  - erythropoietin
  Arms: Multifactorial Intensified therapy
Drug: aspirin — Antiplatelet therapy (in all patients without contraindications):
  - aspirin up to 160 mg/die
  Arms: Multifactorial Intensified therapy

SUMMARY:
The NID-2 study, a multicentric study (21 centres enrolled), was planned in two phases:

Phase 1(observational study, completed in September 2005): after the identification of a type-2 diabetic population with typical Diabetic Nephropathy (DN), to study of the rate of renal and cardiovascular events during a middle term follow-up.

Phase 2(interventional study, started in October 2005): after randomization in two groups, a group (intervention group) is treated with an intensive multifactorial intervention whose aim is to reduce morbidity and mortality due to diabetic complications. The other group (control group) continues the conventional therapy . To avoid bias in the treatment in each center, the randomization was performed for centre.

DETAILED DESCRIPTION:
The same patients that completed the first phase of the NID-2 study (observation) were enrolled for the phase 2 of the study (intervention).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients
* albumin extraction rate (AER= >30 mg/die (micro- or macro-albuminuric ranges) in at least two determinations in the last six months
* diabetic retinopathy
* patients followed in the outpatients clinic for at least 12 months

Exclusion Criteria:

* type 1 diabetic patients
* <40 years old

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinando C Sasso, MD, PhD, Study Director — Università della Campania "Luigi Vanvitelli", Naples, Italy; Roberto Minutolo, MD, MD, Principal Investigator — Università della Campania "Luigi Vanvitelli", Naples, Italy; Luca De Nicola, MD, MD, Study Chair — Università della Campania "Luigi Vanvitelli", Naples, Italy
Locations (1):
- Department of Advanced Medical and Surgical Sciences, Università della Campania "Luigi Vanvitelli", Naples, Italy, Naples, Italy

REFERENCES:
- [Background] Sasso FC, De Nicola L, Carbonara O, Nasti R, Minutolo R, Salvatore T, Conte G, Torella R. Cardiovascular risk factors and disease management in type 2 diabetic patients with diabetic nephropathy. Diabetes Care. 2006 Mar;29(3):498-503. doi: 10.2337/diacare.29.03.06.dc05-1776. PMID 16505495
- [Background] Minutolo R, Sasso FC, Chiodini P, Cianciaruso B, Carbonara O, Zamboli P, Tirino G, Pota A, Torella R, Conte G, De Nicola L. Management of cardiovascular risk factors in advanced type 2 diabetic nephropathy: a comparative analysis in nephrology, diabetology and primary care settings. J Hypertens. 2006 Aug;24(8):1655-61. doi: 10.1097/01.hjh.0000239303.93872.31. PMID 16877970
- [Derived] Sasso FC, Simeon V, Galiero R, Caturano A, De Nicola L, Chiodini P, Rinaldi L, Salvatore T, Lettieri M, Nevola R, Sardu C, Docimo G, Loffredo G, Marfella R, Adinolfi LE, Minutolo R; NID-2 study group Investigators. The number of risk factors not at target is associated with cardiovascular risk in a type 2 diabetic population with albuminuria in primary cardiovascular prevention. Post-hoc analysis of the NID-2 trial. Cardiovasc Diabetol. 2022 Nov 7;21(1):235. doi: 10.1186/s12933-022-01674-7. PMID 36344978
- [Derived] Sasso FC, Pafundi PC, Simeon V, De Nicola L, Chiodini P, Galiero R, Rinaldi L, Nevola R, Salvatore T, Sardu C, Marfella R, Adinolfi LE, Minutolo R; NID-2 Study Group Investigators. Efficacy and durability of multifactorial intervention on mortality and MACEs: a randomized clinical trial in type-2 diabetic kidney disease. Cardiovasc Diabetol. 2021 Jul 16;20(1):145. doi: 10.1186/s12933-021-01343-1. PMID 34271948
- [Derived] Sasso FC, Lascar N, Ascione A, Carbonara O, De Nicola L, Minutolo R, Salvatore T, Rizzo MR, Cirillo P, Paolisso G, Marfella R; NID-2 study group. Moderate-intensity statin therapy seems ineffective in primary cardiovascular prevention in patients with type 2 diabetes complicated by nephropathy. A multicenter prospective 8 years follow up study. Cardiovasc Diabetol. 2016 Oct 13;15(1):147. doi: 10.1186/s12933-016-0463-9. PMID 27733159

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of patients originally enrolled in our study cohort, 538 patients with negative history of cardiovascular events were considered eligible and 111 further added from three new centers. 189 patients from 10 clinics were excluded prior to randomization due to their refusal to participate, 65 individuals due to change of either center or residence
Groups:
- Conventional Therapy: Control group patients will continue their usual therapy. During the study such patients could receive all the therapeutic modifications according to the good medical practice of the specialist.
  current therapy: the patients have to be treated according the standard good medical practice by any center
- Intensified Therapy: Intensive multifactorial intervention is performed to achieve goals for the following risk factors: hypertension, hyperglycaemia, lipids, anaemia. New antihypertensive drugs will be added one by one until achievement of BP target (<130/80 mmHg).
  Therapy for Hypertension
  1. Step1 - irbesartan 300 mg/die and ramipril 10 mg/die
  2. Step 2 (Diuretic) - hydrochlorothiazide 12.5-25 mg/die, if creatinine <2 mg/dL / furosemide 25-75 mg/die, if creatinine ≥2 mg/dL
  3. Step 3 - amlodipine up to 10 mg/die
  4. Step 4 - atenolol up to 100 mg/die
  5. Step 5 - doxazosin up to 4 mg/die
  6. Step 6 - Clonidine
  Therapy for Hyperglycaemia (to achieve HbA1c <7): insulin
  Therapy for hypercholesterolemia (to reduce LDL <100 mg/dl) --> simvastatin till 80 mg/die
  Therapy for hypertriglyceridemia (to reduce triglycerides <150 mg/dl and/or increase HDL >40-50 mg/dl) --> fibrate
  Treatment of anaemia: erythropoietin
  Antiplatelets (all patients without contraindications): aspirin till 160 mg/die
Period: Overall Study
Arm/Group | Conventional Therapy | Intensified Therapy
Started | 188 | 207
Completed | 169 | 199
Not Completed | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Therapy | Intensified Therapy | Total
Number analyzed (Participants) | 188 | 207 | 395
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 104 | 168
  >=65 years | 124 | 103 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.8) | 66.1 (9) | 67.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants] — number and percentage
  Participants
    Female | 105 | 104 | 209
    Male | 83 | 103 | 186
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 188 | 207 | 395

OUTCOME MEASURES:

1. Primary Outcome: "Number of Participants With Overall Fatal and Non-fatal, Major Adverse Cardiovascular Events (MACEs)"
Description: number of MACEs in the two groups are reported. In addition, The primary endpoint was analyzed with event curves for the time-to-first event based on Kaplan-Meier analysis. Cox regression model was used to calculate hazard ratio (HR) and 95% Confidence Interval (CI). Due to the cluster randomized study design, a Cox shared-frailty model was fitted. multivariable model was adjusted for selected potential confounders: age, sex, systolic blood pressure (SBP), hemoglobin, estimated glomerular filtration rate (eGFR), albuminuria, HbA1c, total cholesterol and triglycerides (log-scaled) to reduce risk of bias.
Time Frame: 4 years (in the case the number of events needed by sample size is not reached at the expected 4-year time frame, primary end point will be assessed after the follow-up phase)
Population: number of MACEs reported will be at the end of the whole study period (follow-up) due to the fact that number needed to treat (NNT) at end of intervention was not reached)
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Therapy | Intensified Therapy
Number analyzed (Participants) | 188 | 207
Participants | 146 | 116
Statistical Analysis 1: Comparison: Conventional Therapy vs Intensified Therapy; Test type: Other; p < 0.05, Regression, Cox; Cox Shared Frailty Model, adjusted for age, sex, SBP, Hb, eGFR, albuminuria, HbA1c, total cholesterol, triglycerides (log-scaled) to reduce bias risk; Cox Proportional Hazard = 0.48

2. Secondary Outcome: "Number of Participants Who Achieved of BP, HbA1c and Total, HDL and LDL Cholesterol Goals at the End of Intervention Phase"
Description: Achievement of targets at end of intervention was performed applying generalized estimating equation (GEE) models, further adjusting for baseline values as covariate.
Time Frame: 13 years
Measure: Count of Participants; unit: Participants
Groups:
- Multifactorial Intensified Therapy: An intensive multifactorial intervention according Scientific Guidelines is performed to achieve the goals for the following risk factors: hypertension, hyperglycaemia, lipids, anaemia.
  In particular, new antihypertensive drugs will be added one by one until the achievement of blood pressure target (<130/80 mmHg).
  Therapy for hypertension:
  step 1: irbesartan 300 mg/die and ramipril 10 mg/die Step 2: Diuretic (hydrochlorothiazide 12.5-25 mg/die if serum creatinine <2 mg/dl, furosemide 25-75 mg/die if serum creatinin ≥2 mg/dl) Step 3: amlodipine up to 10 mg/die
Arm/Group | Standard of Care (SoC) Therapy | Multifactorial Intensified Therapy
Number analyzed (Participants) | 169 | 199
Participants | 150 | 191

ADVERSE EVENTS:
Time Frame: up to 13 years
Arm/Group | Conventional Therapy | Intensified Therapy
All-Cause Mortality (participants affected / at risk) | 103/188 | 86/207
Serious Adverse Events (participants affected / at risk) | 88/188 | 69/207
Other Adverse Events (participants affected / at risk) | 5/188 | 8/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Therapy (N=188) | Intensified Therapy (N=207)
Acute Myocardial Infarction (Cardiac disorders) | 44 (44) | 32 (32)
stroke (Cardiac disorders) | 28 (28) | 19 (19)
revascularization (Cardiac disorders) | 13 (13) | 16 (16)
major amputation (General disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Therapy (N=188) | Intensified Therapy (N=207)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) — if fasting glycemia <= 70 mg/dL
Hypotension (General disorders) | 2 (2) | 2 (2) — if systolic blood pressure <= 100 mmHg
End Stage Renal Disease (Renal and urinary disorders) | 2 (2) | 3 (3) — if eGFR (CKD-EPI) < 15 ml/min

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes